CLINICAL TRIAL: NCT01790438
Title: A Comparison of LY2605541 Versus Human Insulin NPH as Basal Insulin Treatment in Insulin-Naïve Patients With Type 2 Diabetes Mellitus Not Adequately Controlled With 2 or More Oral Antihyperglycemic Medications: An Open-Label, Randomized Study
Brief Title: A Study to Compare a New Long-Acting Insulin (LY2605541) and Human Insulin NPH in Participants With Type 2 Diabetes
Acronym: IMAGINE 6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12143; I2R-MC-BIAK (Other: Eli Lilly and Company); 2012-003941-13 (EudraCT Number)
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Results first posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2605541; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2605541 (Experimental): Administered by subcutaneous (SC) injection once daily in the morning or at bedtime. Initial dose is 10 units (or less for some of the participants in Korea) and is adjusted weekly based on Fasting Blood Glucose (FBG). LY2605541 will be given alone or in combination with up to 3 pre-study oral antihyperglycemic medications [OAM(s)] whose use is not excluded in combination with insulin. Treatment may last up to 26 weeks.
  Interventions: Drug: LY2605541; Drug: Oral Antihyperglycemic Medications (OAM)
- Human Insulin NPH (Active Comparator): Administered by SC injection once daily at bedtime. Initial dose is 10 units (or less for some of the participants in Korea) and is adjusted weekly based on FBG. Human insulin NPH will be used alone or in combination with up to 3 pre-study OAM(s) whose use is not excluded in combination with insulin. Treatment may last up to 26 weeks. Some participants who are unable to achieve glycemic control after at least 12 weeks of treatment with a single injection of NPH may be asked to add a second injection prior to the morning meal.
  Interventions: Drug: Human Insulin NPH; Drug: Oral Antihyperglycemic Medications (OAM)

INTERVENTIONS:
Drug: LY2605541
  Arms: LY2605541
Drug: Human Insulin NPH
  Arms: Human Insulin NPH
Drug: Oral Antihyperglycemic Medications (OAM)

SUMMARY:
The purpose of this study is to compare LY2605541 and human insulin isophane suspension (NPH) using the following measures for participants treated for up to 26 weeks:

* Change in participants' overall blood sugar control
* The rate of night time low blood sugar episodes
* The number of participants that reach blood sugar targets without low night time blood sugar episodes
* The total number of low blood sugar episodes reported

ELIGIBILITY:
Inclusion Criteria:

* Have had type 2 diabetes mellitus for at least 1 year, not treated with insulin
* Have been receiving 2 or more OAMs for at least 3 months prior to the study
* Have a hemoglobin A1c (HbA1c) of 7.0% to 11.0%, inclusive, at screening
* Have a body mass index (BMI) less than or equal to 45.0 kilograms per square meter (kg/m^2)
* Women of childbearing potential are not breastfeeding, have a negative pregnancy test at screening and randomization, do not plan to become pregnant during the study, have practiced reliable birth control for at least 6 weeks prior to screening and will continue to do so during the study and until 2 weeks after the last dose of study drug

Exclusion Criteria:

* Have used insulin therapy in the past 2 years (except for use during pregnancy or for short term use for acute conditions)
* Have been treated with glucagon-like peptide-1 (GLP-1) receptor agonist, rosiglitazone, pramlintide, or weight-loss medication within 3 months before screening
* For participants on OAMs: have any restrictions for cardiac, renal, and hepatic diseases in the local product regulations
* Are taking, or have taken within the 90 days before screening, prescription or over-the-counter medications to promote weight loss
* Have had any episodes of severe hypoglycemia, diabetic ketoacidosis, or hyperosmolar state/coma within 6 months prior to screening
* Have cardiac disease with functional status that is New York Heart Association Class III or IV
* Have a history of renal transplantation, or are currently receiving renal dialysis or have serum creatinine greater than or equal to 2 milligrams per deciliter (mg/dL) [177 millimoles per liter (mmol/L)]
* Have obvious clinical signs or symptoms of liver disease [excluding nonalcoholic fatty liver disease (NAFLD)], acute or chronic hepatitis, nonalcoholic steatohepatitis (NASH), or elevated liver enzyme measurements
* Have had a blood transfusion or severe blood loss within 3 months prior to screening or have known hemoglobinopathy, hemolytic anemia, or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the measurement of HbA1c
* Have active or untreated cancer, have been in remission from clinically significant cancer(other than basal cell or squamous cell skin cancer) for less than 5 years, or are at increased risk for developing cancer or a recurrence of cancer in the opinion of the investigator
* Are receiving chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy (excluding topical, intranasal, intraocular, and inhaled preparations) or have received such therapy within the 8 weeks immediately preceding screening
* Have fasting triglycerides greater than 400 mg/dL (4.5 mmol/L) at screening
* Have an irregular sleep/wake cycle (for example, participants who sleep during the day and work during the night) in the investigator's opinion
* Are using or have used any of the following lipid-lowering medications: niacin preparations as a lipid-lowering medication and/or bile acid sequestrants within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern Time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (63):
- United States (20):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tempe, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomfield Hills, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Levittown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
- Canada (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spruce Grove, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burnaby, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. John's, Newfoundland and Labrador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- Czechia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brandýs nad Labem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pardubice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plzen 2-Slovany
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eisenach
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hohenmölsen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saarbrücken
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Ingbert-Oberwürzbach
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schkeuditz
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyöngyös
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagykanizsa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pápa
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
- Puerto Rico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Lomas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yabucoa
- South Korea (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucheon-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sungnam-Si
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teruel

REFERENCES:
- [Derived] Qu Y, White RD, Ruberg SJ. Accurate Collection of Reasons for Treatment Discontinuation to Better Define Estimands in Clinical Trials. Ther Innov Regul Sci. 2023 May;57(3):521-528. doi: 10.1007/s43441-022-00491-0. Epub 2022 Dec 21. PMID 36542287

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2605541: Administered by subcutaneous (SC) injection once daily in the morning or at bedtime. Initial dose was 10 units and was adjusted weekly based on Fasting Blood Glucose (FBG). LY2605541 was given alone or in combination with up to 3 pre-study oral antihyperglycemic medications [OAM(s)] whose use was not excluded in combination with insulin. Treatment may have lasted up to 26 weeks.
- Human Insulin NPH: Administered by SC injection once daily at bedtime. Initial dose was 10 units and was adjusted weekly based on FBG. Human insulin isophane suspension (NPH) was used alone or in combination with up to 3 pre-study OAM(s) whose use was not excluded in combination with insulin. Treatment may have lasted up to 26 weeks. Some participants who were unable to achieve glycemic control after at least 12 weeks of treatment with a single injection of NPH may have been asked to add a second injection prior to the morning meal.
Period: Overall Study
Arm/Group | LY2605541 | Human Insulin NPH
Started | 428 | 213
Received at Least One Dose of Study Drug | 427 | 212
Completed | 393 | 202
Not Completed | 35 | 11
Not completed — Adverse Event | 3 | 2
Not completed — Death | 4 | 0
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 13 | 2
Not completed — Physician Decision | 3 | 1
Not completed — Sponsor Decision | 0 | 3
Not completed — Protocol Required Discontinuation | 7 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- LY2605541: Administered by SC injection once daily in the morning or at bedtime. Initial dose was 10 units and was adjusted weekly based on FBG. LY2605541 was given alone or in combination with up to 3 pre-study OAM(s) whose use was not excluded in combination with insulin. Treatment may have lasted up to 26 weeks.
- Human Insulin NPH: Administered by SC injection once daily at bedtime. Initial dose was 10 units and was adjusted weekly based on FBG. Human insulin NPH was used alone or in combination with up to 3 pre-study OAM(s) whose use was not excluded in combination with insulin. Treatment may have lasted up to 26 weeks. Some participants who were unable to achieve glycemic control after at least 12 weeks of treatment with a single injection of NPH may have been asked to add a second injection prior to the morning meal.
- Total: Total of all reporting groups
Arm/Group | LY2605541 | Human Insulin NPH | Total
Number analyzed (Participants) | 428 | 213 | 641
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.86 (9.76) | 59.79 (10.10) | 59.17 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 107 | 316
  Male | 219 | 106 | 325
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants who were not located in the United States were reported in the "Unknown or Not Reported" category for ethnicity.
  Participants
    Hispanic or Latino | 148 | 73 | 221
    Not Hispanic or Latino | 195 | 105 | 300
    Unknown or Not Reported | 85 | 35 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 53 | 25 | 78
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 9 | 36
  White | 345 | 178 | 523
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 112 | 60 | 172
  Hungary | 24 | 11 | 35
  Czechia | 23 | 12 | 35
  Mexico | 21 | 11 | 32
  Puerto Rico | 46 | 19 | 65
  Canada | 25 | 13 | 38
  Argentina | 31 | 14 | 45
  Poland | 37 | 19 | 56
  Spain | 29 | 16 | 45
  Germany | 30 | 15 | 45
  South Korea | 50 | 23 | 73
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meters (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meters (kg/m^2) | 30.80 (5.57) | 31.04 (5.03) | 30.88 (5.40)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 10.87 (6.46) | 11.40 (7.01) | 11.05 (6.65)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 26 Weeks in Hemoglobin A1c (HbA1c)
Description: Glycosylated hemoglobin A1 (HbA1c) is a test that measures a participant's average blood glucose level over a 2 to 3 month timeframe. Least Squares (LS) means were calculated by mixed model repeated measures (MMRM) using treatment, stratification factors (country, sulfonylureas/meglitinide use [Yes/No]), visit, treatment-by-visit interaction, and baseline HbA1c as the fixed effects.
Time Frame: Baseline, 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 420 | 212
percentage of HbA1c | -1.73 (0.04) | -1.36 (0.06)

2. Secondary Outcome: 30-Day Adjusted Rate of Total and Nocturnal Hypoglycemic Events
Description: Hypoglycemic episodes are defined as an event which is associated with reported signs and symptoms of hypoglycemia, and/or a documented blood glucose (BG) concentration of <=70 milligram per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]). A nocturnal hypoglycemic event is defined as any total hypoglycemia event that occurred between bedtime and waking. Group mean rates of total and nocturnal hypoglycemia (per 30 days) are presented and were calculated from negative binomial regression models with treatment, baseline sulfonylurea/meglitinide use, baseline event rate of the corresponding hypoglycemia as covariates, log (exposure/30 days) as the offset in the model. Group Mean is estimated by taking the inverse link function on individual participant covariates first and then averages over all participants.
Time Frame: Baseline through 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable hypoglycemic data at baseline and with at least one post-baseline value.
Measure: Mean (Standard Error); unit: episodes per participant per 30 days
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 425 | 212
episodes per participant per 30 days
  Total | 1.46 (0.09) | 1.73 (0.13)
  Nocturnal | 0.31 (0.04) | 0.61 (0.07)

3. Secondary Outcome: Percentage of Participants With HbA1c ≤6.5% and <7.0%
Description: Percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100.
Time Frame: 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable HbA1c data.
Measure: Number; unit: Percentage of Participants
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 420 | 212
Percentage of Participants
  HbA1c ≤6.5% | 43.4 | 24.1
  HbA1c <7.0% | 66.3 | 44.7

4. Secondary Outcome: Fasting Serum Glucose (FSG) (by Laboratory)
Description: LS means were calculated from MMRM using treatment, stratification factors (country, sulfonylureas/meglitinide use [Yes/No]), baseline HbA1c strata [≤8.5% or >8.5%]), visit, treatment-by-visit interaction, and baseline value of the response variable as the fixed effects.
Time Frame: 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable FSG.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 422 | 212
milligrams per deciliter (mg/dL) | 112.61 (1.56) | 118.60 (2.20)

5. Secondary Outcome: Fasting Blood Glucose (FBG) (by Self Monitoring)
Description: as for outcome 4
Time Frame: 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable FBG data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 423 | 209
milligrams per deciliter (mg/dL) | 111.37 (1.15) | 109.75 (1.60)

6. Secondary Outcome: 6-Point Self-Monitored Blood Glucose (SMBG)
Description: 6-point SMBG profiles were obtained on 3 nonconsecutive days in the week prior to Weeks 0, 4, 8, 12, 16, and 26. The SMBG measurements were performed while fasting (prior to the morning meal [breakfast]), prior to the midday meal (lunch), prior to the evening meal (dinner), at bedtime, at approximately 0300 hours, and the next day fasting (prior to the morning meal). LS means were calculated by MMRM using treatment, stratification factors (country, sulfonylureas/meglitinide use [Yes/No]), ], baseline HbA1c strata [≤8.5% or >8.5%]), visit, treatment-by-visit interaction, and baseline SMBG at the same time point of the response variable as the fixed effects.
Time Frame: 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable blood glucose data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 400 | 204
mg/dL
  Pre-morning meal: number analyzed (Participants) | 400 | 203
  Pre-morning meal | 111.22 (1.15) | 109.56 (1.61)
  Pre-midday meal: number analyzed (Participants) | 396 | 202
  Pre-midday meal | 123.78 (1.75) | 133.77 (2.44)
  Pre-evening meal: number analyzed (Participants) | 392 | 204
  Pre-evening meal | 130.90 (1.75) | 146.99 (2.41)
  Bedtime: number analyzed (Participants) | 383 | 199
  Bedtime | 144.14 (1.96) | 159.17 (2.72)
  0300 hours: number analyzed (Participants) | 372 | 192
  0300 hours | 116.35 (1.55) | 117.66 (2.15)
  Pre-morning meal the next day | 110.42 (1.18) | 109.03 (1.65)

7. Secondary Outcome: Change From Baseline to 26 Weeks in Body Weight
Description: LS means were calculated by MMRM using treatment, stratification factors (country, sulfonylureas/meglitinide use [Yes/No]), baseline HbA1c strata [≤8.5% or >8.5%]), visit, treatment-by-visit interaction, and baseline weight as the fixed effects.
Time Frame: Baseline, 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 419 | 212
kilograms (kg) | 2.02 (0.16) | 2.34 (0.22)

8. Secondary Outcome: HbA1c
Description: HbA1c is a test that measures a participant's average blood glucose level over a 2 to 3 month timeframe. LS means were calculated by MMRM using treatment, stratification factors (country, sulfonylureas/meglitinide use [Yes/No]), visit, treatment-by-visit interaction, and baseline HbA1c as the fixed effects.
Time Frame: 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 420 | 212
percentage of HbA1c | 6.76 (0.04) | 7.12 (0.06)

9. Secondary Outcome: Insulin Dose Per Kilogram (kg) of Body Weight
Description: LS means were calculated by MMRM using treatment, stratification factors (country, sulfonylureas/meglitinide use [Yes/No]), baseline HbA1c strata [≤8.5% or >8.5%]), visit, and treatment-by-visit interaction as the fixed effects.
Time Frame: 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable insulin dose and body weight data.
Measure: Least Squares Mean (Standard Error); unit: units per kilogram
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 423 | 211
units per kilogram | 0.40 (0.01) | 0.35 (0.02)

10. Secondary Outcome: Time to Steady-State (Stable Maximum Dose)
Description: Steady-state was defined as the first local maximum dose (peak dose value) of LY2605541 or human insulin NPH within the window of -2 to +2 weeks. The median time to steady-state of basal insulin dose estimated from Kaplan-Meier analysis was summarized by treatment.
Time Frame: Baseline through 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable steady state data.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 427 | 212
weeks | 7.14 [6.57 to 8.14] | 5.86 [5.14 to 6.29]

11. Secondary Outcome: Change From Baseline to 26 Weeks in European Quality of Life - 5 Dimension 3 Levels (EQ-5D-3L) Index
Description: The EQ-5D-3L is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a three level scale 1-3 (no problem, some problems, and extreme problems). These combinations of attributes were converted into a weighted health-state Index Score according to the United States (US) population-based algorithm. The EQ-5D-3L US based index scores ranged from -0.11 to 1.0 where a score of 1.0 indicates perfect health. LS means were calculated from ANCOVA using treatment, stratification factor (country, baseline sulfonylurea sulfonylureas/meglitinide use [Yes/No], baseline HbA1c strata [≤8.5% or >8.5%]) and baseline value of EQ-5D-3Las covariates.
Time Frame: Baseline, 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable EQ-5D-3L data. Missing endpoints were imputed with the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 397 | 204
units on a scale | 0.02 (0.01) | 0.01 (0.01)

12. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ) Score
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. The questionnaire measures satisfaction from the following 5 domains: Inconvenience of Regimen, Lifestyle Flexibility, Glycemic Control, Hypoglycemic Control, Insulin Delivery Device. Data presented are the transformed score on a scale of 0-100, higher scores indicate better treatment satisfaction. LS means were calculated using analysis of variance (ANOVA) adjusting for treatment and stratification factors (country, baseline sulfonylureas/meglitinide use [Yes/No], baseline HbA1c [≤8.5% or >8.5%]).
Time Frame: 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable ITSQ data. Missing endpoints were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 419 | 211
units on a scale | 85.04 (0.63) | 83.84 (0.89)

13. Secondary Outcome: Change From Baseline to 26 Weeks in Adult Low Blood Sugar Survey (LBSS) Scores
Description: Adult LBSS (also referenced as Hypoglycemia Fear Survey - II [HFS-II]) contains 33 items, with each item scored on a 5-point response scale: 0 (never) to 4 (always). Items are categorized in 2 domains: Behavior (or avoidance) with 15 items and Worry (or affect) with 18 items. Sum all the items to obtain a total score (range 0-132). Higher total scores reflect greater fear of hypoglycemia. LS means were calculated using analysis of covariance (ANCOVA) adjusting for treatment, stratification factor (country, baseline sulfonylureas/meglitinide use [Yes/No]), baseline HbA1c (≤8.5% or >8.5%), and baseline value of LBSS.
Time Frame: Baseline, 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable LBSS data. Missing endpoints were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 400 | 206
units on a scale | 0.53 (0.72) | 2.05 (1.01)

14. Secondary Outcome: Change From Baseline to 26 Weeks in Lipid Profile
Description: Lipid profile includes total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), and triglycerides. LS means for post-baseline measures were calculated using MMRM with the fixed effects of stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, sulfonylureas/meglitinide use, and LDL-C [<100 mg/dL and ≥100 mg/dL], except for the LDL-C outcome variable), visit, treatment, visit-by-treatment interaction, and baseline value of corresponding lipid outcome variable. LS means for End Of Study measures were calculated using ANCOVA adjusting for stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, sulfonylureas/meglitinide use, and LDL-C [<100 mg/dL and ≥100 mg/dL]except for the LDL-C outcome variable), treatment, and baseline value of corresponding lipid outcome variable.
Time Frame: Baseline, 26 Weeks; Baseline, End Of Study (EOS) (Up to 30 Weeks)
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable lipid data. Missing endpoints for End Of Study measures were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 420 | 212
mg/dL
  Total cholesterol, 26 Weeks | 2.08 (1.42) | 2.86 (2.00)
  Total cholesterol, End Of Study (Up to 30 Weeks) | -0.12 (1.36) | 2.94 (1.92)
  HDL, 26 Weeks | -0.24 (0.31) | 0.41 (0.44)
  HDL, End Of Study (Up to 30 Weeks) | 0.53 (0.31) | 0.40 (0.44)
  LDL, 26 Weeks | 3.01 (1.24) | 5.90 (1.74)
  LDL, End Of Study (Up to 30 Weeks) | 2.54 (1.20) | 3.89 (1.69)
  Triglycerides, 26 Weeks | -1.49 (4.62) | -15.38 (6.49)
  Triglycerides, End Of Study (Up to 30 Weeks) | -20.34 (4.79) | -0.45 (6.74)

15. Secondary Outcome: Percentage of Participants With Insulin Antibodies
Description: The percentage of participants with a positive treatment-emergent anti-LY2605541 antibody response (TEAR) is summarized. TEAR was defined as change from baseline to postbaseline in the anti-LY2605541 antibody level either (1) from undetectable to detectable or (2) from detectable to the value with at least 130% relative increase from baseline. Percentage of participants was calculated by dividing the number of participants with TEAR anytime during the treatment period by the total number of participants analyzed, multiplied by 100.
Time Frame: Baseline to 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable anti-drug (LY2605541) antibodies (ADA) data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 422 | 212
percentage of participants | 19.7 | 45.8

16. Secondary Outcome: Intra-Participant Variability in FBG by Standard Deviation
Description: Glucose variability was assessed by between-day variability as measured by the standard deviation or the coefficient of variation of the FBG of the last 7 days prior to the visit using SMBG. LS means were calculated by MMRM using treatment, stratification factors (country, sulfonylureas/meglitinide use [Yes/No], baseline HbA1c strata [≤8.5% or >8.5%]), visit, treatment-by-visit interaction, and baseline FBG variability as the fixed effects.
Time Frame: 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable FBG data.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 421 | 208
mg/dL | 14.44 (0.50) | 19.07 (0.70)

17. Secondary Outcome: Intra-Participant Variability in FBG by the Coefficient of Variation
Description: Glucose variability was assessed by between-day variability as measured by the standard deviation or the coefficient of variation of the FBG of the last 7 days prior to the visit using SMBG.
Time Frame: 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable FBG data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 421 | 208
mg/dL | 12.87 (0.40) | 17.05 (0.56)

18. Secondary Outcome: Percentage of Participants With Total and Nocturnal Hypoglycemic Events
Description: Hypoglycemic episodes are defined as an event which is associated with reported signs and symptoms of hypoglycemia, and/or a documented blood glucose (BG) concentration of <=70 milligram per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]). A nocturnal hypoglycemic event is defined as any total hypoglycemia event that occurred between bedtime and waking. Percentage of participants was calculated by the number of participants with at least one hypoglycemia divided by the total number of participants analyzed, multiplied by 100.
Time Frame: Baseline through 26 Weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 425 | 212
percentage of participants
  Total | 76.7 | 83.5
  Nocturnal | 41.6 | 67.5

19. Secondary Outcome: Percentage of Participants With HbA1c <7.0% and Without Nocturnal Hypoglycemia
Description: Hypoglycemic episodes are defined as an event which is associated with reported signs and symptoms of hypoglycemia, and/or a documented blood glucose (BG) concentration of <=70 milligram per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]). A nocturnal hypoglycemic event is defined as any total hypoglycemia event that occurred between bedtime and waking. Percentage of participants was calculated by the number of participants reaching target HbA1c without nocturnal hypoglycemia divided by the total number of participants analyzed, multiplied by 100.
Time Frame: 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable HbA1c data and hypoglycemia data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 420 | 212
percentage of participants | 39.1 | 12.6

20. Secondary Outcome: Percentage of Participants With Injection Site Reactions
Description: The percentage of participants with at least one treatment-emergent injection site reaction is presented. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH.
Measure: Number; unit: percentage of participants
Groups:
- LY2605541: Administered by SC injection once daily in the morning or at bedtime. Initial dose is 10 units and is adjusted weekly based on FBG. LY2605541 will be given alone or in combination with up to 3 pre-study OAM(s) whose use is not excluded in combination with insulin. Treatment may last up to 26 weeks.
- Human Insulin NPH: Administered by SC injection once daily at bedtime. Initial dose is 10 units and is adjusted weekly based on FBG. Human insulin NPH will be used alone or in combination with up to 3 pre-study OAM(s) whose use is not excluded in combination with insulin. Treatment may last up to 26 weeks. Some participants who are unable to achieve glycemic control after at least 12 weeks of treatment with a single injection of NPH may be asked to add a second injection prior to the morning meal.
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 427 | 212
percentage of participants | 0.9 | 1.4

21. Secondary Outcome: Rate of Severe Hypoglycemic Events
Description: Hypoglycemic event are defined as an event which is associated with reported signs and symptoms of hypoglycemia, and/or a documented blood glucose (BG) concentration of <=70 milligram per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]). A severe hypoglycemic event was defined as a hypoglycemic episode requiring assistance of another person to actively administer carbohydrates, glucagon, or other resuscitative actions. The hypoglycemia rate per 100 years during a defined period was calculated by the number of hypoglycemia events within the period divided by the number of days participant at risk within the period*36525 days.
Time Frame: Baseline through 26 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: events per 100 participant years
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 425 | 212
events per 100 participant years | 1.00 (0.71) | 0.00 (0.00)

22. Secondary Outcome: Percentage of Participants With Severe Hypoglycemic Events
Description: Hypoglycemic event are defined as an event which is associated with reported signs and symptoms of hypoglycemia, and/or a documented blood glucose (BG) concentration of <=70 milligram per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]). A severe hypoglycemic event was defined as a hypoglycemic episode requiring assistance of another person to actively administer carbohydrates, glucagon, or other resuscitative actions. The percentage of participants with at least one severe hypoglycemia is presented. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 Weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 425 | 212
percentage of participants | 0.5 | 0.0

23. Secondary Outcome: Change From Baseline to 26 Weeks in European Quality of Life (EQ-5D-3L) - Visual Analog Scales (VAS) Scores
Description: The EQ-5D-3L is a generic, multidimensional, health-related, quality-of-life instrument. Overall health state score was self-reported using a visual analogue scale (VAS) marked on a scale of 0 to 100 with 0 representing worst imaginable health state and 100 representing best imaginable health state.
Time Frame: Baseline, 26 Weeks
Population: Participants who received at least one dose of LY2605541 or human insulin NPH with evaluable EuroQol-5D-3L data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2605541 | Human Insulin NPH
Number analyzed (Participants) | 399 | 206
units on a scale | 2.52 (0.68) | 1.41 (0.95)

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug.
Arm/Group | LY2605541 | Human Insulin NPH
Serious Adverse Events (participants affected / at risk) | 28/427 | 9/212
Other Adverse Events (participants affected / at risk) | 228/427 | 111/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2605541 (N=427) | Human Insulin NPH (N=212)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (3)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/209 (0) | 1/107 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (4) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 2 (2) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0/209 (0) | 1/107 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 (N=427) | Human Insulin NPH (N=212)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 13 (16) | 6 (9)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 5 (8)
Nausea (Gastrointestinal disorders) | 6 (6) | 3 (5)
Toothache (Gastrointestinal disorders) | 6 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (3)
Fatigue (General disorders) | 1 (1) | 5 (5)
Oedema peripheral (General disorders) | 11 (14) | 3 (3)
Bronchitis (Infections and infestations) | 8 (8) | 4 (4)
Herpes zoster (Infections and infestations) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 7 (8) | 7 (8)
Nasopharyngitis (Infections and infestations) | 29 (39) | 23 (34)
Sinusitis (Infections and infestations) | 6 (7) | 5 (7)
Tooth infection (Infections and infestations) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 18 (23) | 5 (5)
Urinary tract infection (Infections and infestations) | 10 (14) | 4 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (8) | 2 (2)
Weight increased (Investigations) | 14 (15) | 5 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 8 (10)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (11) | 3 (6)
Dizziness (Nervous system disorders) | 4 (4) | 7 (8)
Headache (Nervous system disorders) | 23 (30) | 9 (17)
Hypoaesthesia (Nervous system disorders) | 6 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 11 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (5)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Hypertension (Vascular disorders) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days